CLINICAL TRIAL: NCT03108469
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of ISIS 546254 for Preventive Treatment of Chronic Migraine
Brief Title: Efficacy and Safety of IONIS-PKKRx for Preventive Treatment of Chronic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Smith, Timothy R., M.D. (Individual)
Collaborators: Clinvest Research, LLC (Industry); Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy Smith, Principal Investigator, Smith, Timothy R., M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-001IS
Record Dates: First submitted 2017-03-27; First posted 2017-04-11 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Chronic Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: At randomization (Visit 2), neither the subject nor the investigator will be aware to which treatment group the subject has been assigned. Investigational product will be drawn and administered in a double blind format. If needed, for safety and proper treatment of the subject, the investigator can unblind the subject's treatment assignment to determine which treatment has been assigned and institute appropriate follow-up care. When possible, Sponsor and Clinvest should be notified prior to unblinding study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IONIS-PKKRx (ISIS 546254) (Active Comparator): Those randomized to IONIS-PKKRx (ISIS 546254) will receive subcutaneous injections containing 1.00 mL (200mg) weekly for weeks 1-16.
  Interventions: Drug: IONIS-PKKRx (ISIS 546254)
- Placebo (Placebo Comparator): Those randomized to placebo will receive subcutaneous injections containing 1.00 mL (200mg) weekly for weeks 1-16.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IONIS-PKKRx (ISIS 546254) — Those randomized to IONIS-PKKRx (ISIS 546254) will receive subcutaneous injections containing 1.00 mL (200mg) of IONIS- PKKRx (ISIS 546254) weekly for weeks 1-16.
  Arms: IONIS-PKKRx (ISIS 546254)
Other: Placebo — Those randomized to placebo will receive subcutaneous injections 1.00 mL (200mg) weekly for weeks 1-16.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and changes in the number of migraine and headache days with repeated subcutaneous administration of IONIS-PKKRx (ISIS 546254) or placebo in subjects with chronic migraine.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multi-center study in subjects with chronic migraine. The study will consist of 7 office visits, 6 Sample collection visits and 3 phone call assessments. Subjects agreeing to participate in the study and meeting the entry criteria assessed at the screening visit, will begin a 28 day baseline period to confirm their diagnosis, and establish a baseline frequency of migraine and headache days. During the baseline period, subjects will continue treating their migraines in their usual manner. They will monitor headache activity, migraine related symptoms, and medication usage with an electronic daily headache diary.

Subjects who, after completing the baseline, continue to meet entrance criteria will be eligible to enter into the 4 month treatment phase. They will be randomized according to the Clinvest generated randomization schedule. A total of 30 randomized subjects will enter the treatment phase receiving IONIS-PKKRx (ISIS 546254; SC) or placebo in a 1:1 design. Study drug or placebo will be administered weekly for 16 weeks. A short phone call to assess any treatment related adverse events will take place 1 and 2 days after randomization. Daily electronic diary assessments will collect headache frequency and severity, associated migraine symptoms, acute medication usage, and the emergence of unusual symptoms and adverse events. Subjects will return to the site at weeks 4, 8, and 12 for investigational product (IP) accountability/dispensing, medication and medication updates, biomarker/lab sample collection, and assessment of adverse events. An end of treatment visit will take place 16 weeks after randomization.

Subjects will have a follow-up safety visit one month after their last dosage of IP ) for assessment of any adverse events (AE) and satisfaction and a final safety phone call 2 months following their last office visit (3 months after last dose of IP) for assessment of any adverse events (AE). Subjects will continue to complete headache diaries through Visit 7. Subjects will also have hematology samples collected every other week starting after Visit 2 through Day 154.

Safety and tolerability will be monitored by the Investigators. Patients who discontinue study treatment prematurely should complete any follow-up visits associated with the most recent dose and should move into and complete the Follow-up Phase.

Subjects will undergo sampling for (pharmacokinetics) PK, coagulation, chemistry, hematology, and optional future biomedical research, as specified in the schedule of procedures.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must meet the following criteria at the screening visit to enter this study:

1. male or female, in otherwise good health, 18 to 65 years of age.
2. history of chronic migraine meeting the diagnostic criteria listed in the International Classification of Headache Disorders (ICHD-III beta version, 2013), as follows:

   a. History of frequent headaches suggestive of chronic migraine (15 or greater days of qualifying headaches per month) for at least three months prior to screening b. Verification of headache frequency through prospectively collected baseline information during the 28-day run-in phase demonstrating headaches on at least 15 days, with at least 8 days per month fulfilling any ONE of the following; i. Qualify as being a migraine attack ii. Relieved by migraine specific acute medications
3. onset of migraine before age 50.
4. stable pattern of migraine pattern for at least 3 months prior to screening.
5. not currently taking a migraine preventive OR has been taking a stable dose of a preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.

   i. Subjects on migraine preventative should have stable headache pattern ii. Injections of onabotulinumtoxinA are allowable if subject has completed at least 2 injection cycles and agrees to maintain a regular injection cycle for the duration of the study

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from entering this study:

1. unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
2. pregnant, actively trying to become pregnant, or breast-feeding.
3. history of medication overuse (MO) of opioids, or butalbital, as defined by ICHD-3 beta criteria and/or MO during baseline period.
4. history of substance abuse and/or dependence, in the opinion of the Investigator.
5. unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Smith, MD, Principal Investigator — Clinvest Research, LLC
Locations (2):
- United States (2):
  - StudyMetrix, City of Saint Peters, Missouri
  - Clinvest Research, LLC, Springfield, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- IONIS-PKKRx (ISIS 546254): Those randomized to IONIS-PKKRx (ISIS 546254) received subcutaneous injections containing 1.00 mL (200mg/mL) weekly for weeks 1-16.
- Placebo: Those randomized to placebo will receive subcutaneous injections containing 1.00 mL weekly for weeks 1-16.
Period: Overall Study
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Started | 15 | 15
Completed | 11 | 11
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (13.04) | 38.4 (10.83) | 37.16 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Migraine Days
Description: Compare the efficacy of ISIS 546254 in the preventive treatment of chronic migraine, measured by the number of monthly migraine days comparing baseline to the final month of the 4-month treatment period for subjects treated with ISIS 546254 vs. placebo.
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Mean (Standard Error); unit: Days
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
Days
  Baseline | 14.267 (1.48) | 14.133 (1.17)
  Treatment Month | 11.067 (2.08) | 9.867 (1.80)

2. Secondary Outcome: Headache Severity
Description: Evaluate the efficacy of ISIS 546254 in the preventive treatment of chronic migraine, measured by the monthly headache severity comparing baseline to the final month of the 4-month treatment period for subjects treated with ISIS 546254 vs. placebo. Headache severity scale ranges from 1 (Mild) to 3 (Severe).
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline | 1.605 (0.106) | 1.538 (0.084)
  Treatment Month | 1.202 (0.146) | 0.994 (0.170)

3. Secondary Outcome: Headache Days
Description: Compare the efficacy of ISIS 546254 in the preventive treatment of chronic migraine, measured by the number of monthly headache days comparing baseline to the final month of the 4-month treatment period for subjects treated with ISIS 546254 vs. placebo.
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Mean (Standard Error); unit: Days
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
Days
  Baseline | 22.267 (1.27) | 23.733 (0.86)
  Treatment Month | 17.733 (2.11) | 14.333 (1.76)

4. Secondary Outcome: Number of Subjects Reporting a ≥ 50% Reduction in the Number of Migraine Headaches
Description: Compare the number of patients meeting 50% response criteria, response defined as a ≥ 50% reduction in the number of headaches from baseline to the final month of the 4-month treatment period for subjects treated with ISIS 546254 vs. placebo.
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 2 | 6

5. Secondary Outcome: Count of Migraine Headache Days Requiring Use of Migraine Medication
Description: Compare the count of the number of headache days requiring use of medication for the treatment of migraine or headache pain (i.e., acute and rescue or breakthrough medication use) from baseline to the final month of the 4-month treatment period for subjects treated with ISIS 546254 vs. placebo.
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Mean (Standard Error); unit: Days
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
Days
  Baseline | 7.2 (1.64) | 14.733 (2.09)
  Treatment Month | 4.733 (1.64) | 7.733 (2.00)

6. Secondary Outcome: Migraine Specific Quality of Life (MSQ) Questionnaire Score
Description: Compare scores from baseline to the final month of the 4-month treatment period in the Migraine Specific Quality of Life (MSQ) Questionnaire for subjects treated with ISIS 546254 vs. placebo.
  The MSQ total score is derived from the summation of fourteen questions on the MSQ. Answer options for the MSQ are coded as: 1 = None of the time, 2 = A little bit of the time, 3 = Some of the time, 4 = A good bit of the time, 5 = Most of the time, 6 = All of the time. The range of total MSQ score for each time point is 14 to 84, with higher scores indicating more effects of migraine on the subject's daily activities.
Time Frame: Comparing baseline to treatment period, up to 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 50.133 (2.40) | 50.133 (2.63)
  Treatment Month | 41.133 (3.46) | 40.733 (3.16)

7. Secondary Outcome: Physician Global Impress of Change (PGIC) Score
Description: Compare the end of treatment month 4 in the physician global impress of change (PGIC) for subjects treated with ISIS 546254 vs. placebo.
  The PGIC is a one item questionnaire asking, "Since the beginning of treatment in this study, how would you describe this patient's change (if any) in their overall status?". The answer option for the PGIC is coded as: 3 = Very Much Improved, 2 = Much Improved, 1 = Minimally Improved, 0 = No Change, -1 = Minimally Worse, -2 = Much Worse, -3 = Very Much Worse, with negative scores indicating the subject's overall status has decreased while in the study and positive scores indicating the subject's overall status has increased while in the study.
Time Frame: Evaluating the treatment period, but collected at the end of treatment, up to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 0.867 (0.215) | 1.00 (0.258)

8. Secondary Outcome: Subject Global Impress of Change (SGIC) Score
Description: Compare the end of treatment month 4 in the subjects' global impression of change (SGIC) for subjects treated with ISIS 546254 vs. placebo.
  The SGIC is a one item questionnaire asking, "Since the beginning of treatment in this study, how would you describe the change (if any) in your overall status?". The answer option for the SGIC is coded as: 3 = Very Much Improved, 2 = Much Improved, 1 = Minimally Improved, 0 = No Change, -1 = Minimally Worse, -2 = Much Worse, -3 = Very Much Worse, with negative scores indicating the subject's overall status has decreased while in the study and positive scores indicating the subject's overall status has increased while in the study.
Time Frame: Evaluating the treatment period, but collected at the end of treatment, up to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 0.867 (0.291) | 1.13 (0.350)

ADVERSE EVENTS:
Time Frame: 196 days
Arm/Group | IONIS-PKKRx (ISIS 546254) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 15/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IONIS-PKKRx (ISIS 546254) (N=15) | Placebo (N=15)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IONIS-PKKRx (ISIS 546254) (N=15) | Placebo (N=15)
Injection site erythema (General disorders) | 15 (96) | 0 (0)
Injection site induration (General disorders) | 9 (31) | 0 (0)
Injection site pain (General disorders) | 11 (51) | 0 (0)
Injection site pruritus (General disorders) | 5 (23) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 0 (0) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03108469/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03108469/SAP_001.pdf